CLINICAL TRIAL: NCT01610089
Title: RDCRN 5110, Nitric Oxide Flux and Ureagenesis in Argininosuccinate Synthetase Deficiency (ASSD)(Citrullinemia I)(Version 24Feb12, NIH Approved 4/5/2012)
Brief Title: Nitric Oxide Flux and Ureagenesis in Argininosuccinate Synthetase Deficiency (ASSD)(Citrullinemia I)
Acronym: NOASSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Brendan Lee, Professor, Molecular and Human Genetics, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: H-27226
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Citrullinemia
Keywords: citrullinemia; argininosuccinate synthetase deficiency; nitric oxide; urea
MeSH Terms: conditions — Citrullinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stable isotope infusion (Experimental): Infusion of isotopes [15N2-ureido] arginine, [5-13C,4, 4, 5, 5-D4] citrulline, [15N]citrulline, 15N sodium nitrate and [15N][18O3] potassium nitrate,[18O][13C]urea.
  Interventions: Other: stable isotope infusion

INTERVENTIONS:
Other: stable isotope infusion — Control subjects: [15N2-ureido] arginine (0.69 mg/kg); [5-13C,4,4,5,5-D4] citrulline (0.18mg/kg); 15N citrulline (0.03mg/kg); 15N sodium nitrate (0.003 mg/kg), [15N][18O3] potassium nitrate (0.03 mg/kg) and [18O][13C]urea (1 mg/kg)over 10 minutes. Followed by a 8-hour infusion of [15N2-ureido] arginine (0.69 mg/kg/hr); [5-13C,4,4,5,5-D4] citrulline (0.18mg/kg/hr), [15N][18O3] potassium nitrate (0.003 mg/kg/hr) and [18O][13C]urea (0.1 mg/kg/hr).
  Citrullinemia type 1 subjects,[15N2-ureido] arginine (4.14 mg/kg); [5-13C,4,4,5,5-D4] citrulline (1.08 mg/kg); 15N citrulline (0.18mg/kg); 15N sodium nitrate (0.003 mg/kg), [15N][18O3] potassium nitrate (0.03 mg/kg) and [18O][13C]urea (1 mg/kg)over 10 minutes, followed by a 8-hour infusion of [15N2-ureido] arginine (4.14 mg/kg/hr); [5-13C,4,4,5,5-D4] citrulline (1.08 mg/kg/hr), [15N][18O3] potassium nitrate (0.003 mg/kg/hr) and [18O][13C]urea (0.1 mg/kg/hr).
  Other Names: stable isotopes

SUMMARY:
The urea cycle consists of a series of chemical reactions through which the body converts toxic waste- nitrogen into a substance called urea that can be disposed of easily. While disposal of nitrogen is the major function of the urea cycle, recent research has shown that some enzymes of the urea cycle are also important for the production of nitric oxide. Nitric oxide is an important chemical that has many functions in the human body including regulation of blood pressure. Through this study, the investigators will study the production of nitric oxide in subjects with citrullinemia type 1 by administering stable isotopes to these subjects. Stable isotopes are harmless compounds that can be used to track and measure the production of specific compounds in the human body. The overall goal of this study is to understand if citrullinemia patients have a deficiency of nitric oxide production. This knowledge may have an impact on the treatment of patients with citrullinemia.

DETAILED DESCRIPTION:
This is an interventional, case control study to investigate the production of nitric oxide in patients with citrullinemia type I. Through the infusion of isotopes [15N2-ureido] arginine, [5-13C,4, 4, 5, 5-D4] citrulline, [15N]citrulline, 15N sodium nitrate and [15N][18O3] potassium nitrate, the flux of citrulline and nitrate through the urea cycle pathway will be measured in conjunction with an independent measure of total plasma arginine flux. This will be informative in dissecting the contributions of de novo production of arginine vs. exogenous contribution of arginine into total body NO flux. Total body urea production will be measured by the isotopic dilution of constantly infused [18O][13C]urea. These flux measurements will be correlated with the level of residual enzyme activity and clinical phenotype in these citrullinemia patients. The investigators plan to enroll three patients with citrullinemia.

Three unaffected control subjects will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be adults (18 years and older) with confirmed diagnosis of Argininosuccinate Synthetase Deficiency (ASSD) (Citrullinemia I) who are able to perform study procedures.
* Diagnosis of citrullinemia I must be confirmed by a >10 fold elevation of citrulline in plasma and/or decreased AS enzyme activity in cultured skin fibroblasts or other appropriate tissue and/or identification of pathogenic mutation in the AS gene.
* Subject must be able to take oral or G-tube medication and have a history of adequate compliance of diet and treatment.
* If a woman of child bearing potential and sexually active, participant agrees to use an acceptable method of birth control.
* Most recent serum creatinine level must be less than or equal to 1.5 mg/dl. Serum creatinine measurement may be performed at the subject's local laboratory, but must have been obtained within one year of enrollment.
* Participant agrees to travel to Baylor College of Medicine for the study.
* Control subjects must be over eighteen years of age with no chronic or acute health issues.

Exclusion Criteria:

* Pregnancy, current acute illness and current hyperammonemic episode.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Flux of citrulline and nitrate through the urea cycle pathway will be measured in conjunction with an independent measure of total plasma arginine flux. | 0, 6, 7 and 7.5 hours of infusion
  Endpoint data to be collected include measurement of isotopic enrichments drawn at 0, 6, 7 and 7.5 hours of infusion. Measurements will include urea, carbon-arginine, guanido-arginine, citrulline, nitric oxide, nitrate and 15N-nitrate.

SECONDARY OUTCOMES:
Total body urea production will be measured by the isotopic dilution of constantly infused [18O][13C]urea. | 0, 6, 7 and 7.5 hours of infusion
  Endpoint data to be collected include measurement of isotopic enrichments drawn at 0, 6, 7 and 7.5 hours of infusion. Measurements will include urea, carbon-arginine, guanido-arginine, citrulline, nitric oxide, nitrate and 15N-nitrate.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Lee, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- See also: Baylor College of Medicine Website — http://www.bcm.edu/